CLINICAL TRIAL: NCT00864409
Title: Local Infiltration Analgesia With Ropivacaine Versus Placebo in Bilateral Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Lasse Andersen, MD, Hvidovre University Hospital
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: KF-01-2006-4062
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Postoperative Pain; Hip Arthroplasty
Keywords: postoperative pain; total hip arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Hip 1 (Active Comparator): high volume local anesthetic infiltration
  Interventions: Drug: ropivacaine 0,2%
- Hip 2 (Placebo Comparator)
  Interventions: Drug: saline.9%

INTERVENTIONS:
Drug: ropivacaine 0,2% — Local wound infiltrtation with 170 mL ropivacaine 2 mg/mL
  Arms: Hip 1
Drug: saline.9% — Wound infiltration with 170 mL sterile saline
  Arms: Hip 2

SUMMARY:
High-volume infiltration analgesia may be effective in postoperative pain management following total hip arthroplasty. In this randomized, double-blind trial patients undergoing bilateral hip arthoplasty are randomized to receive high-volume local anesthetic infiltration in one hip and similar infiltration with saline (placebo) in the other hip.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for bilateral total hip arthroplasty
* able to speak and understand Danish

Exclusion Criteria:

* treatment with opioids or steroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 0-48 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Hviovre University Hospital, Hvidovre, Denmark